CLINICAL TRIAL: NCT04738981
Title: Efficacy and Safety of UC-MSCS for the Treatment of Steroid-resistant aGVHD Following Allo-HSCT: A Multicenter, Randomized, Open-label Trial
Brief Title: Efficacy and Safety of UC-MSCs for the Treatment of Steroid-resistant aGVHD Following Allo-HSCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Southern Medical University, China (Other); Third Military Medical University (Other); Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice president of Peking Univeristy Institute of Hematology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GVHD-PKU2021
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Graft Vs Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — PC61 monoclonal antibody; Basiliximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UC-MSC and anti-CD25 mAb (Experimental): UC-MSC, iv, 1×10^6 cells/kg, once a week, for 4 weeks. Anti-CD25 mAb, iv, 20mg，twice in first week and once a week thereafter, 4 weeks. Other treatment would replace it according to clinical experience if aGVHD continue to progress within 3 weeks of treatment or patients are lack of response after 4 weeks of treatment. The treatment would be repeated in another 4 weeks if patients receive partial response after the first 4 weeks of treatment.
  Interventions: Drug: UC-MSC; Drug: Anti-CD25 mAb
- Anti-CD25 mAb (Active Comparator): Anti-CD25 mAb, iv, 20mg，twice in first week and once a week thereafter, for 4 weeks. Other treatment would replace it according to clinical experience if aGVHD continue to progress within 3 weeks of treatment or patients are lack of response after 4 weeks of treatment. The treatment would be repeated in another 4 weeks if patients receive partial response after first 4 weeks of treatment.
  Interventions: Drug: Anti-CD25 mAb

INTERVENTIONS:
Drug: UC-MSC — UC-MSC, iv, 1×10^6 cells/kg, once a week, for 4 weeks.
  Other Names: Umbilical cord-derived mesenchymal stem cells
  Arms: UC-MSC and anti-CD25 mAb
Drug: Anti-CD25 mAb — Anti-CD25 mAb, iv, 20mg，twice in first week and once a week thereafter, for 4 weeks.
  Other Names: Basiliximab

SUMMARY:
Randomized, open-label, multicenter study to investigate the efficacy and safety of umbilical cord-derived mesenchymal stem cells (UC-MSC) for the treatment of steroid-resistant acute graft-versus-host disease (aGVHD) following allogeneic hematopoietic stem cell transplantation (allo-HSCT), with a view to establishing an effective treatment protocol for steroid-resistant aGVHD.

DETAILED DESCRIPTION:
A total of 130 patients with steroid-resistant aGVHD after allo-HSCT are enrolled in this multicenter, randomized, controlled trial. Patients were randomized to UC-MSC + anti-CD25 monoclonal antibodies (mAb) group and anti-CD25 mAb group. The complete response (CR) rate after 4 weeks of treatment in the two groups will be compared. Adverse events are also recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* 1.Confirmed diagnosed steroid-resistant aGVHD after allo-HSCT. 2. Neutrophile granulocyte (ANC) ≥ 0.5 x 10^9/L. 3. Creatinine below 2 times normal upper limit . 4. Willing and able to sign written informed consent.

Exclusion Criteria:

- 1. Untoleratation of the treatment. 2. Primary disease are not effectively controlled or are progressing. 3. Active infection (Bacteria, fungi, viruses ). 4. Combined with dysfunction of multiple organ. 5. Female patients who are nursing or pregnant, or who contemplate pregnancy during the study period.

6. Patients who are deemed unsuitable for the study by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Rate of complete remission | 4 weeks after treatment
  Complete remission of aGVHD related symptoms and indicators

SECONDARY OUTCOMES:
Overall survival | At the end of Week 4 / 8 / 12 / 24 / 52.
  The time from randomization to death for any reason ( the last follow-up time for missing patients; end date of follow-up for patients who are live at the end of the study).
Rate of partial remission | 4 weeks after treatment
  improvement of aGVHD staging in one or more organs without progression in other organs
Infusion toxicity | From the beginning of to four hours after every infusion of UC-MSC
  Acute toxicity responses include impaired function of heart, kidney and liver

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohui Zhang, doctor, Principal Investigator — Peking University People's Hospital, Peking University Insititute of Hematology
Locations (1):
- Peking University Insititute of Hematology, Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fu H, Sun X, Lin R, Wang Y, Xuan L, Yao H, Zhang Y, Mo X, Lv M, Zheng F, Kong J, Wang F, Yan C, Han T, Chen H, Chen Y, Tang F, Sun Y, Chen Y, Xu L, Liu K, Zhang X, Liu Q, Huang X, Zhang X. Mesenchymal stromal cells plus basiliximab improve the response of steroid-refractory acute graft-versus-host disease as a second-line therapy: a multicentre, randomized, controlled trial. BMC Med. 2024 Feb 27;22(1):85. doi: 10.1186/s12916-024-03275-5. PMID 38413930